CLINICAL TRIAL: NCT01685229
Title: Medical Therapy Versus Balloon Sinus Dilation for Patients With Chronic Rhinosinusitis (MERLOT)
Brief Title: Medical Therapy Versus Balloon Sinus Dilation for Patients With Chronic Rhinosinusitis
Acronym: MERLOT
Status: Completed | Type: Observational
Sponsor: Integra LifeSciences Corporation (Industry)
Collaborators: Acclarent (Industry)
Responsible Party: Sponsor
Other Study IDs: CPR005028
Record Dates: First submitted 2012-09-12; First posted 2012-09-14 (Estimated); Results first posted 2019-05-13 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Sinusitis
MeSH Terms: conditions — Sinusitis | interventions — Practice Management, Medical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Balloon Sinus Dilation: Subjects with chronic sinusitis electing to have a balloon sinus dilation
  Interventions: Device: Balloon sinus dilation
- Medical Management: Subjects with chronic sinusitis electing to continue with medical therapy
  Interventions: Drug: Medical Management

INTERVENTIONS:
Device: Balloon sinus dilation — Subjects electing continued medical therapy group will not have balloon sinus dilation intervention. Subjects electing balloon sinus dilation group will have balloon sinus dilation intervention.
  Other Names: Acclarent Balloon Sinuplasty System
  Groups: Balloon Sinus Dilation
Drug: Medical Management — Subjects who select to continue on medical management rather than have a BSD procedure.
  Groups: Medical Management

SUMMARY:
This post-market study aims to compare health outcomes for Chronic Rhinosinusitis (CRS) patients treated with balloon sinus dilation (BSD) versus continued medical management.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 19 or greater
* Diagnosis of Chronic Rhinosinusitis (CRS)
* Failure of appropriate medical management
* Radiographic evidence of inflammation of the paranasal sinuses
* Surgical candidate
* Willing and able to read and sign the Informed Consent Form and remain compliant with the protocol and study procedures
* Able to read and understand English

Exclusion Criteria:

* Not suitable for balloon dilation for all peripheral sinuses that require treatment
* Clinically significant illness that may interfere with the evaluation of the study
* Patients involved in other clinical studies 30 days prior to study
* Pregnant or lactating females
* Patients unable to adhere to follow-up schedule or protocol requirements

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subjects age 19 or older with radiographically documented CRS
Sampling Method: Non-Probability Sample
Enrollment: 198 (Actual)
Dates: Start 2012-09-01 (Actual); Primary Completion 2015-04-01 (Actual); Study Completion 2015-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Spencer Payne, MD, Principal Investigator — University of Virginia; Christopher Melroy, MD, Principal Investigator — Georgia Nasal and Sinus Institute; Boris Karanfilov, MD, Principal Investigator — Ohio Sinus Institute
Locations (20):
- United States (20):
  - Denver, Colorado
  - Miami, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Savannah, Georgia
  - Vidalia, Georgia
  - Chicago, Illinois
  - Rockford, Illinois
  - South Bend, Indiana
  - Louisville, Kentucky
  - Neptune City, New Jersey
  - Dublin, Ohio
  - Frisco, Texas
  - McKinney, Texas
  - Plano, Texas
  - Charlottesville, Virginia
  - Norfolk, Virginia
  - Richmond, Virginia
  - Beaver Dam, Wisconsin
  - Wauwatosa, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Publication is planned

RESULTS

PARTICIPANT FLOW:
Groups:
- Medical Management: Subjects with chronic sinusitis electing to continue medical therapy
Period: Overall Study
Arm/Group | Balloon Sinus Dilation | Medical Management
Started | 146 | 52
Completed | 120 | 36
Not Completed | 26 | 16
Not completed — Subjects missing Study Exit form | 3 | 1
Not completed — Lost to Follow-up | 16 | 10
Not completed — Withdrawal by Subject | 6 | 5
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Balloon Sinus Dilation | Medical Management | Total
Number analyzed (Participants) | 146 | 52 | 198
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.5 (14.8) | 46.4 (13.3) | 49.4 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 31 | 106
  Male | 71 | 21 | 92

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Change in Chronic Sinusitis Survey (CSS) Score at 24 Weeks Compared to Baseline
Description: The Chronic Sinusitis Survey (CSS) is a 6 question, duration-based survey ("during the past 8 weeks") to evaluate surgical outcomes for CRS patients. The CSS asks three questions each about symptoms and medication usage, yielding a symptom subscore, a medication subscore, and a total score.
  The duration of symptoms is scored 0 ("7-8 Weeks") to 4 ("0 Weeks") and a total score is normalized from 0 (worst) to 100 (best).
  The Primary Endpoint is the comparison of change in total CSS score over 24 weeks for subjects electing BSD versus medical management.
  Change is assessed by using the Mean Change for the CSS total score at 24 weeks compared to baseline. (24-week CSS total score minus Baseline CSS total score).
  Higher score indicates greater improvement.
Time Frame: 24 weeks post treatment
Population: Chronic Sinusitis Survey (CSS) Score Change from Baseline to 24 Weeks for BSD compared to MM
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Balloon Sinus Dilation | Medical Management
Number analyzed (Participants) | 146 | 52
Scores on a scale | 41.9 (23.7) | 27.0 (19.5)

2. Secondary Outcome: Comparison of Change Measured by CSS Medication and Sinusitis Symptom Subscores and Total Score From Baseline
Description: The Chronic Sinusitis Survey (CSS) is a 6 question, duration-based survey ("during the past 8 weeks") used to evaluate surgical outcomes for CRS patients. The CSS asks 3 questions each about symptoms and medication usage, yielding a symptom subscore, a medication subscore, and a total score. The symptom-based section contains pain or pressure, nasal congestion or difficulty to breathe through the nose, and rhinorrhea or postnasal drip. The medication-based section contains: antibiotics, prescription nasal sprays, and sinus medications in pill form. The duration of symptoms is scored 0 ("7-8 Weeks") to 4 ("0 Weeks"), and a total score is normalized from 0 (worst) to 100 (best). The Secondary Endpoint is the comparison of change as measured by average CSS medication and sinusitis symptom sub-scores at 12, 24, and 52 weeks , and average total CSS score at 12 and 52 weeks for subjects electing BSD versus medical management. Higher score indicates greater improvement.
Time Frame: 12, 24, and 52 weeks post treatment
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Balloon Sinus Dilation | Medical Management
Number analyzed (Participants) | 146 | 52
Scores on a scale
  CSS Total Baseline | 28.5 (17.9) | 34.3 (18.4)
  CSS Total Wk 52 | 73.3 (20.2) | 60.2 (22.8)
  CSS Total Wk 52 Change from Baseline | 43.6 (21.7) | 29.9 (20.9)
  CSS Total Wk 12 | 68.7 (20.9) | 56.2 (21.3)
  CSS Total Wk 12 Change from Baseline | 40.6 (22.7) | 21.9 (20.0)
  CSS Symptom Baseline | 21.2 (22.3) | 26.4 (23.3)
  CSS Symptom Wk 12 | 71.0 (25.7) | 56.0 (26.9)
  CSS Symptom Wk 12 Change from Baseline | 50.8 (28.1) | 31.0 (25.3)
  CSS Symptom Wk 24 | 75.1 (24.5) | 60.9 (27.8)
  CSS Symptom WK 24 Change from Baseline | 53.7 (29.9) | 35.2 (31.4)
  CSS Symptom Wk 52 | 74.4 (24.0) | 57.7 (29.1)
  CSS Symptom Wk 52 Change from Baseline | 51.6 (29.4) | 36.4 (29.7)
  CSS Medication Baseline | 35.7 (21.4) | 42.1 (20.2)
  CSS Medication Wk 12 | 66.4 (26.0) | 56.4 (23.3)
  CSS Medication Wk 12 Change from Baseline | 30.5 (27.4) | 12.9 (25.0)
  CSS Medication Wk 24 | 65.6 (25.8) | 61.7 (23.0)
  CSS Medication Wk 24 Change from Baseline | 30.0 (28.8) | 18.8 (21.8)
  CSS Medication Wk 52 | 72.2 (24.8) | 62.7 (27.0)
  CSS Medication Wk 52 Change from Baseline | 35.6 (24.6) | 23.5 (26.1)

3. Secondary Outcome: Change in RSDI
Description: The Rhinosinusitis Disability Index (RSDI) is a 30-question survey which includes 3 individual subscales to measure physical, functional, and emotional scores as well as a total score. There is no specified recall period. Scale values are scored 0 ("Never") to 4 ("Always") and total score ranges from 0 (best) to 120 (worst). Subscores are summed to calculate a total score. Higher score indicates increased impact of sinus disease.
  The Secondary Endpoint is comparison of change in patient-reported QOL as measured by RSDI total, physical, functional, and emotional sub-scores at 12, 24, and 52 weeks compared to baseline for subjects electing BSD versus medical management. Lower score indicates greater improvement (decreased impact of sinus disease).
Time Frame: 12, 24 and 52 weeks post treatment
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Balloon Sinus Dilation | Medical Management
Number analyzed (Participants) | 146 | 52
Scores on a scale
  RSDI Total Baseline | 47.9 (25.3) | 39.5 (19.9)
  RSDI Total Week 12 | 13.0 (17.8) | 26.0 (20.9)
  RSDI Total Week 12 Change from Baseline | -34.7 (24.2) | -14.7 (17.2)
  RSDI Total Week 24 | 11.6 (19.0) | 22.6 (23.2)
  RSDI Total Week 24 Change from Baseline | -36.0 (26.4) | -18.1 (16.8)
  RSDI Total Week 52 | 9.8 (19.1) | 18.7 (20.0)
  RSDI Total Week 52 Change from Baseline | -36.5 (24.9) | -19.9 (19.6)
  RSDI Physical Baseline | 19.4 (9.7) | 16.8 (7.3)
  RSDI Physical Week 12 | 5.4 (7.0) | 11.4 (8.7)
  RSDI Physical Week 12 Change from Baseline | -13.9 (9.4) | -6.0 (7.5)
  RSDI Physical Week 24 | 5.0 (7.7) | 10.1 (9.3)
  RSDI Physical Week 24 Change from Baseline | -14.1 (10.4) | -7.3 (7.1)
  RSDI Physical Week 52 | 4.4 (7.2) | 9.2 (9.7)
  RSDI Physical Week 52 Change from Baseline | -14.3 (9.9) | -7.9 (8.1)
  RSDI Functional Baseline | 14.9 (8.3) | 11.5 (7.0)
  RSDI Functional Week 12 | 4.0 (6.1) | 7.3 (6.6)
  RSDI Functional Week 12 Change from Baseline | -10.9 (8.2) | -4.8 (5.2)
  RSDI Functional Week 24 | 3.5 (6.0) | 6.5 (7.2)
  RSDI Functional Week 24 Change from Baseline | -11.4 (8.5) | -5.4 (5.1)
  RSDI Functional Week 52 | 2.9 (6.2) | 5.4 (5.9)
  RSDI Functional Week 52 Change from Baseline | -11.5 (8.1) | -5.7 (6.7)
  RSDI Emotional Baseline | 13.6 (9.7) | 11.3 (7.6)
  RSDI Emotional Week 12 | 3.7 (5.7) | 7.5 (7.2)
  RSDI Emotional Week 12 Change from Baseline | -9.9 (9.4) | -3.4 (6.1)
  RSDI Emotional Week 24 | 3.1 (6.0) | 5.9 (7.9)
  RSDI Emotional Week 24 Change from Baseline | -10.5 (9.8) | -5.4 (6.7)
  RSDI Emotional Week 52 | 2.5 (6.4) | 4.1 (5.4)
  RSDI Emotional Week 52 Change from Baseline | -10.7 (9.5) | -6.3 (7.0)

4. Secondary Outcome: Change in SNOT-20
Description: The Sino-Nasal Outcome Test (SNOT-20) is a validated questionnaire consisting of 20 symptom-directed questions and quality of life and health utility assessments.
  Scale values range from 0 (No Problem) to 5 (Problem as bad as it can be).
  Lower score indicates greater improvement.
Time Frame: 12 weeks, 24 weeks, 52 weeks post treatment
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Balloon Sinus Dilation | Medical Management
Number analyzed (Participants) | 146 | 52
Scores on a scale
  SNOT-20 Total Baseline | 2.5 (1.0) | 2.4 (0.9)
  SNOT-20 Symptom Week 12 | 0.9 (0.8) | 1.5 (0.9)
  SNOT-20 Symptom Week 12 Change from Baseline | -1.6 (1.1) | -0.9 (1.0)
  SNOT-20 Symptom Week 24 | 0.9 (0.8) | 1.5 (1.0)
  SNOT-20 Symptom Week 24 Change from Baseline | -1.7 (1.1) | -1.0 (1.1)
  SNOT-20 Symptom Week 52 | 0.9 (0.8) | 1.3 (0.9)
  SNOT-20 Symptom Week 52 Change from Baseline | -1.7 (1.2) | -1.2 (1.0)
  SNOT-20 Social-Emotional Baseline | 2.4 (1.2) | 2.3 (1.1)
  SNOT-20 Social-Emotional Week 12 | 0.7 (0.9) | 1.4 (1.0)
  SNOT-20 Social-Emotional Week 12 Change | -1.7 (1.2) | -0.9 (0.9)
  SNOT-20 Social-Emotional Week 24 | 0.8 (1.0) | 1.3 (1.1)
  SNOT-20 Social-Emotional Week 24 Change | -1.6 (1.2) | -1.0 (1.0)
  SNOT-20 Social-Emotional Week 52 | 0.7 (0.9) | 1.0 (0.8)
  SNOT-20 Social-Emotional Week 52 Change | -1.6 (1.4) | -1.3 (1.0)
  SNOT-20 Total Week 12 | 0.8 (0.8) | 1.4 (0.9)
  SNOT-20 Total Week 12 Change from Baseline | -1.6 (1.0) | -0.9 (0.8)
  SNOT-20 Total Week 24 | 0.8 (0.8) | 1.4 (1.0)
  SNOT-20 Total Week 24 Change from Baseline | -1.6 (1.1) | -1.0 (1.0)
  SNOT-20 Total Week 52 | 0.8 (0.8) | 1.2 (0.8)
  SNOT-20 Total Week 52 Change from Baseline | -1.7 (1.2) | -1.2 (0.9)
  SNOT-20 Symptom Baseline | 2.6 (1.0) | 2.6 (0.9)

5. Secondary Outcome: Change in Disease-specific Medication Usage
Time Frame: 12, 24 and 52 weeks post treatment
Measure: Mean (Standard Deviation); unit: Medications
Arm/Group | Balloon Sinus Dilation | Medical Management
Number analyzed (Participants) | 146 | 52
Medications
  Oral Antibiotics Baseline | 28.1 (15.4) | 22.8 (6.1)
  Oral Antibiotics Week 12 | 5.7 (8.4) | 6.6 (9.5)
  Oral Antibiotics Week 12 Change from Baseline | -22.2 (17.0) | -16.7 (11.4)
  Oral Antibiotics Week 24 | 2.3 (6.6) | 2.8 (6.7)
  Oral Antibiotics Week 24 Change from Baseline | -25.9 (15.8) | -20.5 (10.1)
  Oral Antibiotics Week 52 | 2.0 (5.9) | 1.8 (5.5)
  Oral Antibiotics Week 52 Change from Baseline | -25.8 (15.5) | -22.4 (8.5)
  Oral Steroids Baseline | 7.9 (10.4) | 8.4 (10.0)
  Oral Steroids Week 12 | 3.0 (9.8) | 2.6 (7.0)
  Oral Steroids Week 12 Change from Baseline | -4.9 (13.7) | -6.5 (10.6)
  Oral Steroids Week 24 | 0.8 (3.6) | 0.7 (2.8)
  Oral Steroids Week 24 Change from Baseline | -6.5 (9.9) | -7.9 (9.3)
  Oral Steroids Week 52 | 2.5 (13.9) | 2.6 (9.1)
  Oral Steroids Week 52 Change from Baseline | -4.5 (17.0) | -6.4 (14.4)
  Nasal Steroid Spray Baseline | 53.0 (29.6) | 47.2 (28.1)
  Nasal Steroid Spray Week 12 | 39.7 (40.3) | 69.1 (35.5)
  Nasal Steroid Spray Week 12 Change from Baseline | -13.3 (44.2) | 21.1 (44.1)
  Nasal Steroid Spray Week 24 | 44.6 (42.6) | 66.0 (35.5)
  Nasal Steroid Spray Week 24 Change from Baseline | -9.1 (46.6) | 18.4 (45.5)
  Nasal Steroid Spray Week 52 | 34.8 (41.1) | 57.0 (39.7)
  Nasal Steroid Spray Week 52 Change from Baseline | -17.5 (46.0) | 10.0 (52.1)

6. Secondary Outcome: Missed Days Work/School
Time Frame: 12, 24 and 52 weeks post treatment
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Balloon Sinus Dilation | Medical Management
Number analyzed (Participants) | 146 | 52
Days
  Baseline | 3.0 (9.2) | 1.4 (2.4)
  Wk 24 | 0.2 (0.8) | 0.0 (0.0)
  Wk 52 | 0.4 (2.9) | 0.1 (0.4)
  Wk 24 Change from Baseline | -2.0 (4.4) | -1.3 (2.2)
  Wk 52 Change from Baseline | -1.5 (3.9) | -1.2 (2.2)

7. Secondary Outcome: Number of Sinus-related Medical Care Visits
Time Frame: 12 weeks, 24 weeks, 52 weeks post treatment
Measure: Mean (Standard Deviation); unit: Visits
Arm/Group | Balloon Sinus Dilation | Medical Management
Number analyzed (Participants) | 146 | 52
Visits
  Sinus-Related Visits at Baseline | 2.0 (2.1) | 1.2 (1.6)
  Sinus-Related Visits through 12 weeks | 0.1 (0.3) | 0.1 (0.5)
  Sinus-Related Visits through 24 weeks | 0.1 (0.4) | 0.1 (0.6)
  Sinus-Related Visits through 52 weeks | 0.2 (0.5) | 0.1 (0.6)

8. Secondary Outcome: Number of Sinus Infections
Time Frame: 24 and 52 weeks
Measure: Mean (Standard Deviation); unit: Sinus infections
Arm/Group | Balloon Sinus Dilation | Medical Management
Number analyzed (Participants) | 146 | 52
Sinus infections
  Sinus Infections through 24 weeks | 0.3 (0.6) | 0.3 (0.6)
  Sinus Infections through 52 weeks | 0.5 (0.8) | 0.6 (0.8)

9. Secondary Outcome: Number of Subjects Requiring Revision for Subjects Electing BSD
Description: A revision is defined as an endoscopic sinus surgery procedure on sinuses successfully dilated during index (BSD) procedure due to documented worsening of condition related to those sinuses after the index (BSD) procedure.
Time Frame: 52 weeks
Measure: Number; unit: Participants
Arm/Group | Balloon Sinus Dilation | Medical Management
Number analyzed (Participants) | 146 | 52
Participants | 3 | 0

10. Secondary Outcome: Number of Medical Management Subjects Electing to Cross-over to Balloon Sinus Dilation Procedure
Time Frame: 52 weeks
Measure: Number; unit: Participants
Arm/Group | Medical Management
Number analyzed (Participants) | 52
Participants | 12

11. Secondary Outcome: Post-operative Return to Normal Activity (RTNA)
Time Frame: 2 weeks post treatment
Measure: Mean (Standard Deviation); unit: Days
Groups:
- In-Office: BSD subjects treated in an office setting
- Operating Room: BSD subjects treating in an Operating Room venue
Arm/Group | Balloon Sinus Dilation | In-Office | Operating Room
Number analyzed (Participants) | 146 | 105 | 41
Days | 3.6 (4.1) | 2.8 (3.7) | 5.9 (4.1)

ADVERSE EVENTS:
Description: No AEs were related to the device
Arm/Group | Balloon Sinus Dilation | Medical Management
All-Cause Mortality (participants affected / at risk) | 1/146 | 0/52
Serious Adverse Events (participants affected / at risk) | 6/146 | 0/52
Other Adverse Events (participants affected / at risk) | 49/146 | 8/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Balloon Sinus Dilation (N=146) | Medical Management (N=52)
GI Bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0)
Pancreatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Neuropenic Shock (Immune system disorders) | 1 (1) | 0 (0)
Cancer, Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Bells Palsy, TIA (Nervous system disorders) | 2 (2) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Balloon Sinus Dilation (N=146) | Medical Management (N=52)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 3 (3)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 30 (38) | 4 (4)
URI (Respiratory, thoracic and mediastinal disorders) | 12 (14) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days